CLINICAL TRIAL: NCT03536078
Title: Home Phototherapy for Term Newborns With Icterus, a Clinical Randomized Blinded Trial
Brief Title: Home Phototherapy for Term Newborns With Icterus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 209715
Record Dates: First submitted 2018-03-23; First posted 2018-05-24 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2019-09

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: home phototherapy; parental bonding
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Group allocation blinded to the investigator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phototherapy at hospital (No Intervention): Newborns with icterus that receive treatment while being admitted to hospital.
- Home phototherapy (Experimental): Newborns with icterus receiving phototherapy at home.
  Interventions: Other: home phototherapy

INTERVENTIONS:
Other: home phototherapy
  Arms: Home phototherapy

SUMMARY:
The study is designed as a randomised controlled multicenter study.The primary aim is to investigate if home phototherapy improves parent-child bonding compared to if treatment is performed at the hospital. The investigators will also istudy how home phototherapy is perceived by the parents, impact on breastfeeding and parents stress levels, if the method can be implemented etc.

Patients are included at 5 hospitals in Sweden. The plan is to include 250 term newborns with neonatal icterus at a level that needs phototherapy treatment.

DETAILED DESCRIPTION:
Background: Almost half of all newborns develops jaundice, due to elevated levels of bilirubin. If levels are high phototherapy is needed to reduce the levels of bilirubin. Presently most children with neonatal jaundice in Sweden receives phototherapy admitted to hospital. There is fiberoptic equipment available that can be used at home to treat the newborns.

Aim: Primary aim is to investigate if parent-child bonding is improved with home phototherapy compared to phototherapy performed at the hospital.

Method:The study is designed as a randomised controlled multicenter study. Eligible parents and newborns are randomised to either treatment at home or at the hospital. Demographic data about the newborn such as for example apgar score, gender, time of birth etc are registered. At time of discharge parents answers questionnaires such as for example the Postpartum Bonding Questionnaire (PBQ), the Edinburgh Postnatal Depression Scale (EDPS), the Swedish Parenthood Stress Questionnaire etc. Parents experiences from home phototherapy will also be investigated through semistructured interviews.

Parents will asked to answer questionnaires at the time of discharge as well as at 4-months after discharge.

Analysis of data will be performed by using conventional parametric and non-parametric statistical methods.

The results of the study will be reported as scientific articles and as part of a thesis.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age w36-42.
* Age of newborn 48 hours or more.
* Level of bilirubin 300-400 µmol/l

Exclusion Criteria:

* Immunisation. Bilirubin >400 µmol/l. Asphyxia. Ongoing infection, weightloss > 10%, other severe disease, parents who don´t speak Swedish, parents that are not expected to be able to handle the home phototherapy equipment

Min Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Change in parent-child bonding | Change from discharge to 4-months after discharge
  Measured by parents answering the Postpartum Bonding questionnaire. Score range 0-125, higher is worse.

SECONDARY OUTCOMES:
Change in parents emotional status | Change from discharge to 4 months after discharge
  Measured by parents answering the Edinburgh Postnatal DepressionScale (EDPS). Score range 0-30, higher is worse.
Change in health-related Life quality | Change from discharge to 4 months after discharge
  Measured by parents answering SF-36 (Short Form Health Survey). Score range 36-108, higher is worse.
Change in mothers experience of breastfeeding | Change from discharge to 4 months after discharge
  Measured by mothers answering Maternal Breastfeeding Evaluation Scale.(MBES). Score range 30-150, higher is better.
Parental stress | at 4 months after discharge
  Measured by parents answering the Swedish Parenthood Stress Questionnaire. Score range 34-170, higher is worse.
Transcutaneous bilirubin measurement, and how it is affected by phototherapy | measurements are performed from date of randomization until discharge, assessed up to 4 weeks of age.
  Transcutaneous bilirubin is measured every time a blood sample for bilirubin is checked. The transcutaneous measurements are performed on skin exposed to phototherapy(sternum) and non-exposed skin (sacrum).

CONTACTS AND LOCATIONS:
Overall Officials: Mats Eriksson, Professor, Principal Investigator — Örebro university, Region Orebro County
Locations (5):
- Sweden (5):
  - Childrens department University hospital in Örebro, Örebro, Region Orebro County
  - Childrens department at Mälarsjukhuset/hospital, Eskilstuna
  - Childrens department Falun hospital, Falun
  - Childrens department Halmstad hospital, Halmstad
  - Childrens department Karlstad hospital, Karlstad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pettersson M, Ryen L, Eriksson M, Ohlin A. The cost-effectiveness of home phototherapy for hyperbilirubinemia in neonates: results from a randomized controlled trial. Sci Rep. 2023 Jul 3;13(1):10727. doi: 10.1038/s41598-023-37684-y. PMID 37400561
- [Derived] Pettersson M, Eriksson M, Blomberg K. Parental experiences of home phototherapy for neonatal hyperbilirubinemia. J Child Health Care. 2023 Dec;27(4):562-573. doi: 10.1177/13674935221082404. Epub 2022 Mar 26. PMID 35341337
- [Derived] Pettersson M, Eriksson M, Albinsson E, Ohlin A. Home phototherapy for hyperbilirubinemia in term neonates-an unblinded multicentre randomized controlled trial. Eur J Pediatr. 2021 May;180(5):1603-1610. doi: 10.1007/s00431-021-03932-4. Epub 2021 Jan 19. PMID 33469713